CLINICAL TRIAL: NCT07194018
Title: Evaluation of the Use of Cannabis Oil in Patients With Fibromyalgia
Brief Title: Use of Cannabis Oil in Fibromyalgia
Acronym: FIBRO-CB
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.TerD.24.01
Record Dates: First submitted 2025-08-20; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia; Pain Management; Cannabis; Retrospective Studies
MeSH Terms: conditions — Fibromyalgia; Agnosia; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Use of cannabis oil — Use of cannabis oil on pain relief in patients suffering from fibromyalgia syndrome

SUMMARY:
Recently, medical cannabis has been shown to be effective in chronic pain conditions such as osteoarthritis, neuropathic pain, and other chronic non-cancer pain.

A study showed that fibromyalgia patients who use cannabis report significant improvement in pain symptoms and quality of life. Patients reported a 50% reduction in pain, and many also reported improvements in sleep and overall well-being. Further research found that the use of medical cannabis among patients with fibromyalgia led to significant improvements in pain, sleep quality, and overall quality of life. This study emphasized that adverse effects were generally mild and tolerable. Furthermore, the systematic review by Fitz et al. concluded that cannabis may be effective in treating fibromyalgia, with preliminary evidence indicating improvements in pain and sleep disturbances. However, it also highlighted the need for further randomized controlled trials to confirm these findings and determine how the cannabinoid system interacts with the pain pathway.

Considering that medical cannabis is effective in treating a variety of symptoms, including pain, cachexia and wasting, sleep disorders, severe or persistent muscle spasms, reduced fatigue in multiple sclerosis, chemotherapy-induced nausea, convulsive disorders, post-traumatic stress disorder, and other conditions in palliative and end-of-life care; with this study, given the premises of the effects of medical cannabis, the aim is to analyze its use also in chronic pain as the main symptom of fibromyalgia syndrome.

DETAILED DESCRIPTION:
Fibromyalgia syndrome, also known simply as "fibromyalgia," is a central sensitization syndrome characterized by dysfunction of the neurocircuits responsible for the perception, transmission, and processing of nociceptive afferents, with pain predominantly manifested in the musculoskeletal system.

The link between pathophysiology and treatment is still very weak, and significant efforts are still needed to offer patients treatment targeted at the biological causes of the disease.

To date, the treatment of fibromyalgia is aimed at reducing the main symptoms and must be individualized and multidisciplinary, involving both non-pharmacological measures and, in most patients, drug therapy.

Cannabinoids or cannabinols are chemicals that share the ability to interact with cannabinoid receptors and can be of three types: endocannabinoids, synthetic cannabinoids, and phytocannabinoids.The Company Therapeutic Handbook (PTA) from the hospital pharmacy of the AOU "SS Antonio e Biagio e Cesare Arrigo" in Alessandria provides for the use of cannabis oil from September 2022. Considering that medical cannabis is effective in treating multiple symptoms, including pain, cachexia and wasting, sleep disorders, severe or persistent muscle spasms, and others, this study aims to analyze its use in chronic pain as the main symptom of fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent;
* age ≥ 21 years;
* diagnosis of FM according to the 2016 American College of Rheumatology (ACR) diagnostic criteria;
* failure of previous therapies.

Exclusion Criteria:

* psychiatric disorders,
* history of drug or alcohol addiction,
* fatty liver disease or severe liver disease,
* severe cardiopulmonary disease,
* severe renal failure,
* pregnancy or breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 21 years who have been diagnosed with fibromyalgia according to the 2016 American College of Rheumatology (ACR) diagnostic criteria and who have failed previous therapies.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-10-19 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Through study completion, an average of 1 year
  Scale Numeric Pain Rating Scale (NRS) for pain assessment from 0 (no pain) to 10 (maximum pain)

SECONDARY OUTCOMES:
Number of adverse events | Through study completion, an average of 1 year
  Assess the number of adverse events
Severity of adverse events | Through study completion, an average of 1 year
  Assess the severity of adverse events
Adherence to therapy | Every day through study completion, an average of 1 year
  Assessment of medication intake in the indicated doses and times (patient is "adherent" if they take at least 80% of the prescribed doses , "partially adherent" if they take between 20% and 80%, and "non-adherent" if they take less than 20%).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No